CLINICAL TRIAL: NCT03756181
Title: A Mixed Methods Evaluation Study of Brief Mindfulness-based Stress Reduction and Brief
Brief Title: Mindfulness and Self-Compassion in McGill University
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: issue with project feasibility
Sponsor: Lady Davis Institute (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Soham Rej MD, MSc, Assistant Professor, Dept. of Psychiatrist, McGill University, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A00-B21-18A
Record Dates: First submitted 2018-09-17; First posted 2018-11-28 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Five-week MSC program (MSC5wk) (Experimental): This program adaptation will consist of conducted meditative practices, discussions, and background information within a group setting of no more than 25 students per group. The facilitator may discuss the student's experience and encourage group sharing within the course of the session. These discussions will reinforce the guiding principles of compassion: self-kindness, mindfulness, and common humanity, and will work on soothing the processes of self-criticism, self-neglect and perfectionism that are believed to withhold upon experiencing psychological distress. There will also be sessions dedicated to incorporating self-compassion in daily life, with more detailed instructions, as well as encouraging a 30- minute daily home practice.
  Interventions: Behavioral: Five-week MSC program (MSC5wk)
- Five-week Mindfulness-based Stress Reduction program (MBSR5wk) (Active Comparator): This program adaptation will consist of conducted meditative practices, discussions, and background information within a group setting of no more than 25 students per group. The facilitator will perform a brief check-in and may discuss the student's experience within the course of the session. These discussions will reinforce the guiding principles of meditation: awareness, non-judgment and acceptance and will work on automatic mental processes that are believed to be at the root of experiencing psychological distress. There will also be sessions dedicated to incorporating mindfulness into daily life, with more detailed instructions, as well as encouraging a 30- minute daily home practice.
  Interventions: Behavioral: Five-week MSC program (MSC5wk)

INTERVENTIONS:
Behavioral: Five-week MSC program (MSC5wk) — This program adaptation will consist of conducted meditative practices, discussions, and background information within a group setting of no more than 25 students per group. The facilitator may discuss the student's experience and encourage group sharing within the course of the session. These discussions will reinforce the guiding principles of mindfulness meditation. There will also be sessions dedicated to incorporating or mindfulness in daily life, with more detailed instructions, as well as encouraging a 30- minute daily home practice.
  Other Names: Five-week Mindfulness-based Stress Reduction program (MBSR5wk)

SUMMARY:
Mental health issues are increasingly costly in Quebec. Given most psychological disorders occur before age 24, university-based interventions are appealing to prevent and treat mental illness, especially as rates of psychological distress have peaked among university students in our province. This at-risk population may benefit from new university-based programs, as academic institutions now face limited staffing and an increasing number of students seeking services. Mindfulness-based Stress Reduction (MBSR) programs are a promising approach, reporting substantial increases in emotional regulation. Novel mindful self-compassion (MSC) programs additionally display increasing improvements in resilience, that could foster stronger well-being in highly competitive academic contexts. A few high-quality scientific studies have investigated the impact of university setting MSC programs, but it remains unclear to determine whether MBSR or MSC may be useful in Canadian student populations experiencing psychological distress. This study will rigorously evaluate both programs efficacy and will be the first one to understand the student's experience in both groups.

DETAILED DESCRIPTION:
In Canada, 42 billion dollars are spent per year treating mental health issues. Given that 53% Canadians undergo postsecondary education, the mental health of university students is of great concern, especially as they experience higher proportions of psychological distress ("stress") compared to the general population. Reports indicate a 42.2% of stress levels in university students, which not only poses a significant impact in their academic performance, but also meaningfully contributes to decreased rates of students completing their studies, and in high rates of long-term maladjustment mental illness including depression (15-30%), and anxiety (32.2%). University students are also prone to develop eating disorders (6%), attention-deficit/hyperactivity disorder (4%), post-traumatic stress disorders (3%), drug/substance abuse (2.1%) , and sleep disturbances (5% to 73%).

As the onset of most psychological disorders occurs at age 24, university students may greatly benefit from mental health assistance provided by academic institutions. At McGill University, high rates of psychological distress are experienced by both undergraduate and graduate students, as observed by concerning rates of suicidality (10% of students have considered attempting suicide while at University), trauma (5 to 16%), and testimonials of experiencing social anxiety (61-65 %) and academic distress (55-66%). Moreover, a steady increase in students seeking mental health or counseling services and the increased complexity and severity of symptoms have placed significant attention in the development of strategies addressing university students' psychological well-being.

Implementation science: mental health care in university settings. Many public-sector services systems and provider organizations are in some phase of learning about or implementing evidence-based interventions. Universities represent an optimal setting for reaching young adults with mental health promotion and prevention programs as they are a captive audience, thus reducing adherence problems known to diminish the impact and outcomes of public health interventions in general.

Successful program implementation (i.e., examining the barriers and facilitators of program adherence to an evidence-based program) is directly associated with better outcomes and a translational promise to accelerate knowledge into practice. Efforts to enhance and improve outcome involves ameliorating concordance with evidence-based clinical practice guidelines. However, guidelines for the treatment of mental illnesses are underdeveloped and not routinely well implemented in mental health care, despite the number of evidence-based practices on the rise.

Moreover, studies have found that young people in need of mental health care services show less adherence to prevention and treatment programs, despite the availability of evidence-based practices. In the context of university students, it appears that university students face not only high academic demands and perceived and self-stigmatizing attitudes towards mental illness, but also report limited accessibility (time, transport, and cost) to participate in or adhere to mental health care. Other barriers are related to confidentiality and trust, concern about the characteristics of the provider, difficulty or an unwillingness to express emotion, preferring other sources of help (i.e., family, friends), and worrying about effects on career. In this vein, it remains crucial to systematically study what factors impact program adherence (i.e., attendance on three out of five sessions), and home practice (i.e., continued home practice). Studies also need to understand further how students experience stress and explain the comparative experiences of students participating in different mental health promotion and prevention strategies.

Current treatments in Canada and at McGill: Some studies suggest that approximately 50% of university students experience significant stress (i.e., a reaction observed in the form of depression and anxiety). It is therefore recommended that universities employ preventative interventions that impact large numbers of students (i.e., group-based interventions) instead of merely relying on individual services to meet student needs. Current treatments for psychological distress offered at Canadian universities include health promotion and accessibility, counseling, and medical services. These are limited by lack of coordination, financial constraints, adequate staffing, and primarily reactive response to focus on problems as they arise.

In McGill University, student's support services include the Peer-Support Centre (PSC), counseling services and psychiatric consultation for more severe cases. At the therapeutic level, counseling services offer vocational and therapeutic workshops, therapeutic groups (i.e., Cognitive Behavioral Therapy and Acceptance and Commitment Therapy), and one-on-one counseling services. However, the current wait-time for students with mental health issues to initially meet a counselor and receive urgent support (i.e., being placed on a therapeutic group) is approximately four weeks. This creates significant pressure for McGill Student Services to offer rapid open-access services to students experiencing stress. In this vein, Student Services not only tackles a student's need for support but also actively engages them in mental health prevention promoting continued well-being. Newer "third wave" programs including mindfulness and compassion-based (i.e., Mindful Self-Compassion) interventions are a promising approach, especially as they have gain popularity in educational settings.

Self-compassion interventions: While some research groups have begun evaluating the use of mindfulness programs in university settings (i.e., MBSR), most studies address populations of medical students rather than overall university-level populations. Yet, novel self-compassion programs remain to be examined. While mindfulness-based interventions focus on the non-judgmental experience of the present moment, compassion-based approaches focus on kindly addressing the suffering experience of the experiencer itself. In light with this, compassion-based approaches foreground cultivating compassion towards self and others, given high levels of self-criticism associated with many mental disorders. Compassion greatly benefits mental health and emotional regulation, improves interpersonal and social relations and is considered a significant predictor of well-being and resilience. Novel programs include Mindful Self-Compassion (MSC) which demonstrates solid endurance and resilience effects, and may theoretically have a more significant impact on university students compared to well-known third wave interventions, such as MBSR.

It is relevant to delineate that MBSR's loving-kindness meditation is different from compassion and self-compassion meditation. In loving kindness, the aim is to develop an affective state of unconditional kindness to all people. In compassion, the aim is to cultivate deep and genuine sympathy for those stricken by misfortune and to develop an earnest wish to ease suffering. In self-compassion, the aim is to soothe and comfort the 'self' when any distressing experience arise, remembering that such experiences are part of being human. In this vein, loving kindness is best explained as our attention for all being to be happy, whereas compassion refers to our attention for all beings (or ourselves, in self-compassion) to be free from suffering.

Recently, studies have addressed self-compassion as a moderator of perfectionism and depression in both adolescence and adulthood suggesting that self-compassion interventions may be useful in determining the effects of maladaptive perfectionism. It also appears that self-kindness and mindfulness serve as a buffer of stress as students claim to receive social support and that self-compassion training has an essential impact on measures of depression, anxiety, general well-being, self-compassion, mindfulness, life satisfaction, social connectedness, optimism, self-efﬁcacy, and rumination. Additionally, self-compassionate students are less afraid of failure and are more likely to train again when they fail, have less academic worry and also have a greater sense of self-efficacy. This portrays the student's ability to handle social and academic struggles more effectively, report less depression and homesickness, as well as more satisfaction about their choice of study while at the university.

Limitations to self-compassion interventions: effectiveness and implementation science. To our knowledge, the only study that has examined the effect of MSC in university students was a brief version of MSC compared to a time management intervention in 51 college females. Findings from this study include significantly more significant gains in self-compassion (21%), mindfulness, optimism, self-efficacy and decreases in rumination, strongly suggesting that short versions of MSC may have a substantial potential to improve psychological well-being and resilience of university students. Results from this study, also include medium to high effect size for self-compassion (r=1.19), mindfulness-awareness without judgement (r=0.70), mindfulness-non-reactivity to inner experience (r= 1.20), optimism (r=0.66), self-efficacy (r=0.52), and rumination (r=0.70). Although these effect size measures are of importance, the sample was too small to further determine the effects of the program and interestingly, necessary measures of psychological and vocational influence (both crucial to academic success) were not thoroughly addressed. Furthermore, there are no studies examining impact factors of program implementation (i.e., those associated to student's participation of self-compassion programs), despite a growing interest in implementation science in the educational setting and mental health prevention field. In this study, we will address the issues above to better examine the comparative effectiveness of MSC to MBSR.

Using a mixed methods approach, including a randomized controlled trial and an in-depth qualitative interview, this study will assess the comparative efficacy of newly developed brief Mindful Self-Compassion (MSC) and Mindfulness-based Stress Reduction (MBSR) programs on improving stress in university students. Factors impact group adherence (retention and home practice) will also be explored. Participant's experience of stress and the comparative experience of students participating in both groups will be explained.

ELIGIBILITY:
Inclusion Criteria:

* McGill University Students (Graduate or Undergraduate Students) enrolled or seeking services within McGill Counselling and Mental Health Services
* Age 18 years or older
* Students should have sufficient hearing (or assistive devices) to hear verbal instructions and discussion
* Have an adequate understanding of English and/or French

Exclusion Criteria:

* • Depression (PHQ9) and anxiety (GAD7) ≥12
* Acute psychotic symptoms
* Severe personality problems that will interfere with their ability to function in a group setting
* Acute Suicidal ideation/intent

  * Student scoring ≥12 on either scale will be immediately referred to therapeutic services offered on campus

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress | Change in PSS from 0 to 5-weeks (baseline to post-1).
  The Perceived Stress Scale (Cohen, Kamarck, & Mermelstein, 1983; Cohen et al., 1994) is a standardized,10 item self-report questionnaire used to determine the extent to which a person perceives her or his life to be stressful, by taping experiences of distress related to "how unpredictable, uncontrollable, and overloaded respondents ﬁnd their lives" (Shapiro, Brown, Thoresen, & Plante, 2011). A sample question is "How often have you found that you could not cope with all the things that you had to do?" Participants responded on a 5-point scale ranging from 1 (never) to 5 (very often). Internal consistency reliability was α = .92.

SECONDARY OUTCOMES:
Self-compassion | Change in SCS from 0 to 5-weeks (baseline to post-1).
  The 12-item short form of the Self-Compassion Scale (Raes et al., 2011), assesses the positive and negative aspects of the three main components of self-compassion: Self-Kindness versus Self-Judgment; Common Humanity versus Isolation; and Mindfulness versus Over-Identification (Neff, 2003). Responses are given on a 7-point scale ranging from 1 (almost never) to 7 (almost always). It has good psychometric properties, with high internal consistency and a nearly perfect correlation with the long form of the Self Compassion Scale (Raes et al., 2011). Higher scores correspond to higher levels of self-compassion. Internal reliability is α = .85.
Mindfulness | Change in FFMQ from 0 to 5-weeks (baseline to post-1).
  The Five Facets Mindfulness Questionnaire - Short (Bohlmeijer, ten Klooster, Fledderus, Veehof, & Baer, 2011) is derived from the 39 item Five Facets Mindfulness Questionnaire (Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006). Mindfulness can be conceptualized as a multifaceted construct consisting of five related dimensions: Observing, Describing, Acting with Awareness, Non-judging of Inner Experience, and Non-reactivity to Inner Experience. There are 15 items in this scale, and it is rated on a 5-point Likert scale, ranging from 1 (never or very rarely true) to 5 (very often or always true). In addition to considering scores on the five sub-scales individually, facet scores can be combined to produce an overall mindfulness score. Internal consistency is α = .85 (Baer, Carmody, & Hunsinger, 2012).
Perceived Stress | Change in PSS will be assessed from 0 to 10-weeks (baseline to post-2).
  The Perceived Stress Scale (Cohen, Kamarck, & Mermelstein, 1983; Cohen et al., 1994) is a standardized,10 item self-report questionnaire used to determine the extent to which a person perceives her or his life to be stressful, by taping experiences of distress related to "how unpredictable, uncontrollable, and overloaded respondents ﬁnd their lives" (Shapiro, Brown, Thoresen, & Plante, 2011). A sample question is "How often have you found that you could not cope with all the things that you had to do?" Participants responded on a 5-point scale ranging from 1 (never) to 5 (very often). Internal consistency reliability was α = .92.
Perceived Stress | Change in PSS will be assessed from 5 to 10-weeks (post-1 to post-2).
  The Perceived Stress Scale (Cohen, Kamarck, & Mermelstein, 1983; Cohen et al., 1994) is a standardized,10 item self-report questionnaire used to determine the extent to which a person perceives her or his life to be stressful, by taping experiences of distress related to "how unpredictable, uncontrollable, and overloaded respondents ﬁnd their lives" (Shapiro, Brown, Thoresen, & Plante, 2011). A sample question is "How often have you found that you could not cope with all the things that you had to do?" Participants responded on a 5-point scale ranging from 1 (never) to 5 (very often). Internal consistency reliability was α = .92.
Depression | Change in PHQ-9 from 0 to 5-weeks (baseline to post-1).
  The Patient Health Questionnaire (PHQ-9) (Kroenke & Spitzer, 2002) represents a self-reported 9-item depression scale, and it is based on the DSM-IV criteria for major depressive disorder with responses to questions ranging from 0 ("not at all") to 3 ("nearly every day") for each item. Summed scores ≥10 are considered clinically significant.
Anxiety | Change in GAD-7 from 0 to 5-weeks (baseline to post-1).
  The General Anxiety Disorder-7 (GAD- 7) (Spitzer et al., 2006) is a 7-item tool to measure the severity of various signs of generalized anxiety disorder on a 0 ("not at all") to 3 ("nearly every day") scale. Summed scores ≥10 are considered clinically significant.
Rumination | Change in RRS from 0 to 5-weeks (baseline to post-1).
  The Ruminative Response Scale-NL-Extended (Raes et al., 2003) measures the extent to which they experience ruminative responses when feeling sad or depressed. The scale comprises 26 items with a 4-point response format ranging from 1 (almost never) to 4 (almost always). For the current study, we looked at the brooding subscale that has been identified by (Treynor, Gonzalez, & Nolen-Hoeksema, 2003). Sample items from the five-item brooding subscale include "Why do I have problems other people don't have?" and "Why can't I handle things better?" Reliability of the scale in the present sample was α = .93.
Perfectionism | Change in APS-R from 0 to 5-weeks (baseline to post-1).
  The revised Almost Perfect Scale (APS-R) (Slaney & Ashby, 1996) is a widely used measure of perfectionism. This scale has 23 self-report items and consists of three subscales: Standards (7 items), Discrepancy (12 items), and Order (4 items). Items are responded by using a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree) (Slaney, Rice, Mobley, Trippi, & Ashby, 2001). Reliability estimates have been reported in the moderate to high range. While two of the scales (reflecting high standards and an appreciation of order) measure adaptive perfectionism, a third scale (discrepancy) measures maladaptive perfectionism. Internal consistency has been reported from mid-range to low range (Vandiver & Worrell, 2002).
Connectedness | Change in SCS from 0 to 5-weeks (baseline to post-1).
  The Social Connectedness Scale-Revised (Lee et al., 2001) comprises 20 items and measures the degree of interpersonal closeness that individuals feel with other people, both friends, and society. Sample items include "I feel disconnected from the world around me." Responses were given on a 6-point scale ranging from 1 (strongly agree) to 6 (strongly disagree), with higher scores corresponding to a stronger sense of belonging. The scale has been shown to have good test-retest and internal reliability. Internal reliability in the present study was α = .91.
Optimism | Change in LOT-R from 0 to 5-weeks (baseline to post-1).
  The Life Orientation Test-Revised (LOT-R) is used to measure levels of dispositional optimism (Scheier et al., 1994). The LOT-R comprises 10 items assessing the extent to which individuals expect favorable outcomes for the future (e.g., "I'm always optimistic about my future"). Of the 10 items, three are positively phrased, three are negatively phrased, and four are filler items. Responses are given on a 5-point Likert scale ranging from 0 (strongly agree) to 4 (strongly disagree). After reverse scoring the three negatively phrased items, a total LOT-R score can be calculated by adding scores of all items. Higher scores correspond with higher levels of optimism. The LOT-R has been shown to have good psychometric properties. Reliability of the scale in the present sample was α = .73.
Self-efficacy | Change in SES from 0 to 5-weeks (baseline to post-1).
  The General Self-Efficacy scale (Schwarzer & Jerusalem, 2010), is used to measure participants' beliefs in their ability to deal with potentially challenging situations. It comprises 10 statements (e.g., "I am confident that I could deal efficiently with unexpected events"), rated on a 4-point scale ranging from 1 (not at all true) to 4 (exactly true). Reliability of the scale in the present sample was α = .81.

OTHER OUTCOMES:
Home mindfulness or self-compassion practice | Each week throughout the intervention (weeks 1 through 5)
  Home mindfulness practice will be assessed using weekly homework logs (Baer et al., 2012). Participants will be asked to record the number of minutes of daily home practice of the formal meditation practices taught in either mindfulness or self-compassion programs. They will be also asked to rate from 1 to 5 the degree to which they felt they had followed the mindfulness or self-compassion instructions (1 = not at all, 5 = very much). The instruction will be made clear so that they are not being asked whether they felt it was a "good" practice session, but the degree to which they felt they followed the instructions.
Fidelity of implementation (FOI) | Each week throughout the intervention (weeks 1 through 5)
  At the end of each session, facilitators will be asked to complete a FOI checklist based on the commonly agreed-upon dimensions of fidelity (Dane & Schneider, 1998; Dusenbury, Brannigan, Falco, & Hansen, 2003). A 'comments' section will inquire about future recommendations. We will use an online self-report of FOI similar to the used in C.-Y. S. Lee et al. (2008) that is more related to measuring the facilitator's adherence rather than competence.
Participant's experience of stress | post-1 (at week-5)
  In depth interviews using the MINI (Groleau et al., 2006). The MINI provides an overall structure and sequence of questions, but interviewers must improvise additional questions and probes to clarify responses. Like any open-ended form of interviewing the MINI depends on the interviewer's understanding of the underlying research questions and the broader conceptual framework guiding the inquiry. The MINI allows for the exploration of diverse meanings and ways or reasoning held by interviewees about their experience of stress, whether contradictory or complementary. The MINI guides a conversation that produces narratives that can be used to study individual experience meanings, modes of reasoning, historical sequences, and the sociocultural contexts of experience. In this study, we will evaluate all sections of the MINI (Groleau, Young, & Kirmayer, 2006) which have been modified to address participant's experience of stress and the comparative effects of participating in both groups.
Participant's experience in the groups | post-1 (at week-5)
  In depth interviews using the MINI (Groleau et al., 2006). The MINI provides an overall structure and sequence of questions, but interviewers must improvise additional questions and probes to clarify responses. Like any open-ended form of interviewing the MINI depends on the interviewer's understanding of the underlying research questions and the broader conceptual framework guiding the inquiry. The MINI allows for the exploration of diverse meanings and ways or reasoning held by interviewees about their experience of stress, whether contradictory or complementary. The MINI guides a conversation that produces narratives that can be used to study individual experience meanings, modes of reasoning, historical sequences, and the sociocultural contexts of experience. In this study, we will evaluate all sections of the MINI (Groleau, Young, & Kirmayer, 2006) which have been modified to address participant's experience of stress and the comparative effects of participating in both groups.
Adverse events | Each week throughout the intervention (weeks 1 through 5)
  Given the importance of participant's safety in compassion-based and mindfulness-based programs, a question on adverse events (Dobkin et al., 2012) will be collected weekly and at program end, week-5. These measures may be reported in our manuscripts.

IPD SHARING:
Plan to Share IPD: No